CLINICAL TRIAL: NCT01765855
Title: AN OPEN-LABEL, SINGLE-DOSE, MASS-BALANCE STUDY TO ASSESS THE DISPOSITION OF 14C-LABELED PRT054021 IN HEALTHY MALE SUBJECTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06-005
Record Dates: First submitted 2012-12-28; First posted 2013-01-10 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Health Volunteers
Keywords: Betrixaban; Healthy; Mass Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Oral Betrixaban (Experimental)
  Interventions: Drug: Betrixaban single oral dose

INTERVENTIONS:
Drug: Betrixaban single oral dose

SUMMARY:
This is a open label, single center, single oral dose, study of PRT054021, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men ages of 19 and 55 years old, inclusive
* weighs at least 132 lbs

Exclusion Criteria:

* Clinically significant comorbid disease
* History of substance abuse
* Hemoglobin less than 12.0 g/dl

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
mean (max, tmax, AUC) | Over 336 hours

SECONDARY OUTCOMES:
Percent dose recovered in urine and feces | Over 336 hours